CLINICAL TRIAL: NCT05409781
Title: Prevalence of May-Thurner Syndrome in 1st-degree Relatives of Symptomatic Patients
Acronym: MTS
Status: Withdrawn | Type: Observational
Why Stopped: Decided amongst research group that this project is not feasible
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, Research Nurse Manager, University Hospital of Limerick
Other Study IDs: DVS002
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: May-Thurner Syndrome
MeSH Terms: conditions — May-Thurner Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The aim is to assess the prevalence of May-Thurner syndrome in 1st-degree relatives of previously identified symptomatic patients.

DETAILED DESCRIPTION:
May-Thurner syndrome (MTS) is a condition characterised by compression of the left common iliac vein by the right common iliac artery and the anterior spine of the 5th lumbar vertebrae. Previously thought to be a rare condition, the prevalence of MTS is thought to be underreported. MTS can lead to significant morbidity in the form of chronic venous insufficiency, venous ulceration, lower limb swelling, venous claudication, deep-vein thrombosis, varicose veins, pelvic congestion syndrome, chronic pelvic pain and chronic post-thrombotic syndrome. It is a known risk factor for development of venous incompetence and varicose veins in adolescents and young adults. Furthermore, it is known to be an a causative factor in the development of "unprovoked" DVT in younger patients, however data on the risk of development of DVT in MTS patients has to date, been unavailable.

The pathogenesis of MTS is largely unknown and whilst the condition is known to be more prevalent in females, familial risk factors are largely unknown. To date, no studies have previously assessed the prevalence of MTS in relatives of those with the condition.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, first degree relative with symptomatic May-Thurner syndrome

Exclusion Criteria:

* Those who not give informed consent to be contacted or to be scanned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pathogenesis of MTS is largely unknown and whilst the condition is known to be more prevalent in females, familial risk factors are largely unknown. To our knowledge, no studies have previously assessed the prevalence of MTS in relatives of those with the condition.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence Assessment | 1 year
  To assess the prevalence of May-Thurner syndrome amongst 1st-degree relatives of symptomatic individuals referred to the Vascular Department, University Hospital Limerick using duplex ultrasound imaging

SECONDARY OUTCOMES:
Venous Competence Assessment | 1 year
  To assess concomitant venous incompetence of the lower limb

IPD SHARING:
Plan to Share IPD: No
Np plan to share IPD